CLINICAL TRIAL: NCT04623632
Title: Effect of the Modified Surgeon Assisted Bilateral TAP Block on Time Required for First Analgesic Dose After Cesarean Section Under Spinal Anesthesia:A Randomized,Placebo-controlled, Double Blinded Clinical Trial
Brief Title: Effect of TAP Block on Time Required for First Analgesic Dose After Cesarean Cection Under Spinal Anesthesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Elmaraghy, Lecturer of obstetrics and gynecology - faculty of medicine - Ainshams university, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3
Record Dates: First submitted 2020-11-05; First posted 2020-11-10 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine (Active Comparator): the landmark is at the level of umbilicus 8 to 10 cms from midline bilaterally. A tiny nick is made in the skin with a 18G sharp needle to obliterate the cushion effect. Then an 18 G Tuohy needle will be insert perpendicular to skin directing the needle slightly towards the ipsilateral anterior superior iliac spine just before the closure of peritoneum. After feeling 2 pops of external and internal oblique aponeurosis the drug will be injected after aspiration. The injectate syringes will be prepared under aseptic technique; syringes contained bupivacaine 0.25% 40 ml. Once the plane is reached the surgeon places his hand inside the abdominal cavity at the level of needle insertion to reconfirm needle placement. A bleb is palpated by the surgeon as the injection continues. The back flow of drug after injection is one of the signs that drug has been deposited in the TAP plane
  Interventions: Drug: Transversus abdominus plane block
- Placebo (Placebo Comparator): the landmark is at the level of umbilicus 8 to 10 cms from midline bilaterally. A tiny nick is made in the skin with a 18G sharp needle to obliterate the cushion effect. Then an 18 G Tuohy needle will be insert perpendicular to skin directing the needle slightly towards the ipsilateral anterior superior iliac spine just before the closure of peritoneum. After feeling 2 pops of external and internal oblique aponeurosis the drug will be injected after aspiration. The injectate syringes will be prepared under aseptic technique syringes contained either normal saline 40 ml. Once the plane is reached the surgeon places his hand inside the abdominal cavity at the level of needle insertion to reconfirm needle placement. A bleb is palpated by the surgeon as the injection continues. The back flow of drug after injection is one of the signs that drug has been deposited in the TAP plane
  Interventions: Drug: Transversus abdominus plane placebo

INTERVENTIONS:
Drug: Transversus abdominus plane block — transversus abdominus plane block using 40 ml of bupivacaine 0.25%
  Other Names: Regional analgesia
  Arms: Bupivacaine
Drug: Transversus abdominus plane placebo — injection of 40 ml of normal saline in the transversus abdominus plane
  Arms: Placebo

SUMMARY:
While opioids are the mainstay for post-operative analgesia after caesarean section, they are associated with various side effects. Ultrasound guided transversusabdominis plane (TAP) block has been postulated to provide effective analgesia for caesarean section. However a new technique in TAP block is described which can be used safely by a beginner without any fear of complication whichwill help in providing good postoperative analgesia to maximumnumber of patients.

This study will evaluate the analgesic efficacy of TAP block using Modified Surgeon Assisted Bilateral TAP block for post caesarean analgesia in a randomized controlled trial.

DETAILED DESCRIPTION:
Acute severe pain after cesarean delivery is frequent. At least 10 to 15% of the women develop chronic pain .Effective postoperative analgesia after caesarean section is important because it enables early ambulation and facilitates breast-feeding.

The administration of opioids, local blocks and other analgesic medication is instituted to decrease the duration and intensity of postoperative pain as a part of a multimodal analgesic regimen. The transversusabdominis plane (TAP) block is a regional analgesic technique which blocks T6-L1 nerve branches and has an evolving role in postoperative analgesia for lower abdominal surgeries .

In postoperative analgesia, efficacy of TAP block is equivalent to morphine with the additional benefits of increasing duration of analgesia, reducing postoperative opioid usage, with satisfactory pain relief and few side effects.

The TAP block avoids the risk of neuraxial complications and opioid complications in all patients. TAP block the neural afferents of theanterior abdominal wall after spreading of the local anesthetic agent in the neurofascial plan between the internal oblique and transversusabdominis muscle.

TAP block has been underutilized in spite of having very low complication and high success rate using ultrasound technique This may be due to the lack of availability of ultrasound at most of the centers, lack of training in ultrasound guided block technique.

A new technique can be used in TAP block without the fear of complications in the blind landmark based approach.The advantage of this technique includes avoiding missing the second pop in obese and pregnant patients due to thinning of the internal obliqueaponeurosis, reposition of the needle by surgeon if one enters the peritoneal cavity accidentally. Also there are nil chances of visceral injury thus can be safely used by a beginner without any fear of complication. However, there might be a chance of needle stick injury to the surgeon's hand.

This study aims to evaluate effect of the Modified Surgeon Assisted Bilateral TAP block on time required for first analgesic dose after Cesarean Section under spinal anesthesia

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) class I-II
2. Normal singleton pregnancy.
3. With a gestational age of completed 37 weeks or more.
4. Category ІV cesarean section

Exclusion Criteria:

1. Under the age of 18 or older than 40 years.
2. Obese patients with a BMI >40.
3. ASA III or ASA IV risk groups
4. Patients with contraindications to spinal anesthesia or history of allergy to bupivacaine.
5. patients who received analgesics in the past 24 hours
6. Infection in the region where the block would be performed.
7. Category І- Ц- Ш cesarean section
8. Refusal to participate in the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Time to the first opioid analgesic request | First 24hours after cesarean section
  when will the patient ask for opioid analgesia after cesarean section

SECONDARY OUTCOMES:
Total analgesic requirements in 24 hours Total opioid analgesic requirements in 24 hours | first 24hours after cesarean section
  The number of patients requiring rescue analgesia and the frequency of this analgesia and total analgesic usage will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Adel Shafik, MD, Study Director — AinShams university
Locations (1):
- AinShams university maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Ahmad M, Furqan A, Adnan M, Waris S and Yousuf M (2019):
- [Background] Canakci E, Gultekin A, Cebeci Z, Hanedan B, Kilinc A. The Analgesic Efficacy of Transverse Abdominis Plane Block versus Epidural Block after Caesarean Delivery: Which One Is Effective? TAP Block? Epidural Block? Pain Res Manag. 2018 Oct 17;2018:3562701. doi: 10.1155/2018/3562701. eCollection 2018. PMID 30416635
- [Background] Blanco R, Ansari T, Girgis E. Quadratus lumborum block for postoperative pain after caesarean section: A randomised controlled trial. Eur J Anaesthesiol. 2015 Nov;32(11):812-8. doi: 10.1097/EJA.0000000000000299. PMID 26225500
- [Background] McMorrow RC, Ni Mhuircheartaigh RJ, Ahmed KA, Aslani A, Ng SC, Conrick-Martin I, Dowling JJ, Gaffney A, Loughrey JP, McCaul CL. Comparison of transversus abdominis plane block vs spinal morphine for pain relief after Caesarean section. Br J Anaesth. 2011 May;106(5):706-12. doi: 10.1093/bja/aer061. PMID 21498494
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Background] 6. Roy R and Pattnaik S (2016):
- [Background] 7. Sriramka B, Sahoo N and Panigrahi S (2012):